CLINICAL TRIAL: NCT02419170
Title: Mature Dendritic Cell Vaccination Against Unique Immunogenic Peptides in Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator who manufactured the vaccine left the university.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-x043
Record Dates: First submitted 2015-02-04; First posted 2015-04-17 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma, Non-Small-Cell-Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Component Removal; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery/Apheresis/Cyclophosphamide/Vaccine (Experimental): * Standard of care surgery
  * Apheresis (between Day -28 and Day -7) approximately 12 weeks after surgery
  * Cyclophosphamide 300 mg/m^2 intravenously (Day -4)
  * Personalized vaccine (Day 1)
  * Booster dose of personalized vaccine (Day 43)
  * Booster dose of personalized vaccine (Day 85)
  Interventions: Procedure: Standard of care surgery; Procedure: Apheresis; Drug: Cyclophosphamide; Biological: Personalized mature dendritic cell vaccine

INTERVENTIONS:
Procedure: Standard of care surgery
Procedure: Apheresis
Drug: Cyclophosphamide
  Other Names: Cytoxan®
Biological: Personalized mature dendritic cell vaccine

SUMMARY:
The purpose of this research study is to study the safety and immune response of people who receive a personalized dendritic cell vaccine with the intention of stimulating the immune system to react to lung cancer cells.

DETAILED DESCRIPTION:
Tumor vaccines represent a promising area of clinical investigation in solid tumors based on evidence of clinical activity and minimal toxicity. The underlying hypothesis of this research is that immunization against tumor neoantigens is effectively required to elicit antigen-reactive T cells capable of recognizing and eliminating cancer. Moreover, both quantitative and qualitative improvements in CD8 immunity are necessary (but not sufficient) for clinical response and improved survival. The goal of this study is to build on our prior clinical trial results in melanoma by studying the immune response to tumor neoantigens in patients with stage 1 NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with completely resected stage I non-small cell lung cancer who are not considered for adjuvant post operative therapy.
* Age ≥ 18 years.
* ECOG performance status 0-1.
* HLA-A2 positive.
* Required initial laboratory values (submitted within 14 days prior to registration):

  * WBC > 3,000/mm3
  * Hg ≥ 9.0 gm/dL
  * Platelets >75,000/mm3
  * Serum bilirubin < 2.0 mg/dL
  * Serum creatinine < 2.0 mg/dL
* Sexually active women of childbearing potential must use effective birth control during the trial and for at least two months following the trial, and sexually active men must be willing to avoid fathering a new child while receiving therapy.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Prior treatment with cytotoxic chemotherapy
* Prior treatment with targeted therapy or immunotherapy.
* Active untreated CNS metastasis.
* Active infection.
* Prior malignancy (except non-melanoma skin cancer) within 3 years.
* Pregnant or nursing.
* Concurrent treatment with systemic corticosteroids; local (inhaled or topical) steroids are permitted.
* Known allergy to eggs.
* Prior history or uveitis or autoimmune inflammatory eye disease.
* Known positivity for hepatitis B sAg, hepatitis C antibody, or HIV antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Immunological response as measured by increased numbers of peptide specific CD8+ T cells as calculated by the tetramer assay | 1 year
  -Blood for immunological response is drawn every week from Dose #1 to 6 weeks after Dose #3 (Day 1 to Day 126 = Week 18 and then every 4 weeks until Day 365)
Safety and tolerability of vaccine as measured by adverse events experienced and graded by NCI CTCAE Version 4.0 | 30 days after last vaccine (approximately Day 115)
  Safety will be closely monitored after vaccination. Patients will be observed for 2 hours after the first dose and vital signs recorded every 30 minutes during that time period beginning at the start of the infusion. For each dose thereafter, patients will be observed in the treatment area for 30 minutes after the infusion. The following parameters will be assessed:
  * Local signs and symptoms
  * Systemic signs and symptoms
  * Laboratory evaluations
  * Adverse and serious adverse events
  * Toxicity will be graded according to the NCI's CTCAE version 4.0.

SECONDARY OUTCOMES:
Time to progression (TTP) | 5 years
  These patients have been completed resected so there is no tumor response to monitor. CT scans evaluating for progression will be performed at baseline, following the third vaccine dose, and as per routine care during follow-up (generally every 3 months for the first year and every 6 months for the next 4 years thereafter).

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu